CLINICAL TRIAL: NCT05608382
Title: Effect of an Antiseptic Solution on the Skin Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovation and Research Organization (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SGW2022
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Skin Diseases, Infectious
MeSH Terms: conditions — Skin Diseases, Infectious

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sterile Phosphate Buffer Saline (PBS) (Placebo Comparator)
  Interventions: Other: sterile Phosphate Buffer Saline
- SGW13 (Experimental)
  Interventions: Other: SGW13

INTERVENTIONS:
Other: sterile Phosphate Buffer Saline — control group
  Arms: sterile Phosphate Buffer Saline (PBS)
Other: SGW13 — active comparator
  Arms: SGW13

SUMMARY:
The objective of this study is simulate the clinical use of an antiseptic solution in a 24 hour window and the recovery to baseline conditions at 1 month following application. Efficacy will be simulated as the capacity of the material to reduce or clear the skin bacterial population from a representative skin area: the anteromedial forearm.

ELIGIBILITY:
Inclusion Criteria:

A subject may be eligible for study participation if all of the following criteria are met:

1. Subject is male or female greater than 18 years of age.
2. Subject does not have a history of skin allergies/atopia (e.g. atopic dermatitis).
3. Subject does not have a history of skin disease (e.g scleroderma, vitiligo, psoriasis) or a chronic systemic disease affecting the skin (e.g systemic lupus erythematosus).
4. Subject is willing to have materials applied and follow the protocol.
5. Subject agrees to avoid exposure of the test sites to the sun, chemical product, clothes and to refrain from touching the area of application (for T0 [baseline], T1 [5 minutes], T2 [2 hours]).
6. Subject agrees to refrain from getting a bath/shower before T3 (24 h).
7. Subject agrees to avoid scrubbing, applying, and/or washing the test area with new soap, moistures, powders, lotions, cosmetic or toiletry products during the study.
8. Subject is able to follow directions as outlined in the protocol and anticipates being available for all study visits.
9. Subject is willing to participate in all study evaluations.
10. Subject is in generally good health.
11. Subject is willing to sign the Informed Consent form prior to study participation

Exclusion Criteria:

1. Female subject is pregnant, nursing, planning a pregnancy, or not using adequate birth control.
2. Subject is immunologically compromised or has received specific topical treatment (antimicrobial or not-antimicrobial), during the last month.
3. Subject reports a history of allergies to antiseptics.
4. Subject is currently taking certain medications which, in the opinion of the Principal Investigator, may interfere with the study.
5. Subject has known allergies to skin treatment products or cosmetics, toiletries, and/or topical drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Colony Forming Unit (CFU) count | 5 minutes
  Comparison of the number of CFUs counted for each treatment arm
Colony Forming Unit (CFU) count | 2 hours
  Comparison of the number of CFUs counted for each treatment arm
Colony Forming Unit (CFU) count | 24 hours
  Comparison of the number of CFUs counted for each treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Javad Parvizi, MD, Principal Investigator — Center for Innovation and Research Organization
Locations (1):
- Center for Innovation and Research Organization, Philadelphia, Pennsylvania, United States